CLINICAL TRIAL: NCT05297357
Title: Complementary Weaning With Adult Food Typical of the Mediterranean Diet and it Effect on Taste Development and Eating Habits of Children
Brief Title: Complementary Weaning With Adult Food Typical of the Mediterranean Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Dario Bruzzese, Full Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 213
Record Dates: First submitted 2022-03-12; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Weaning
Keywords: Complementary feeding; Mediterranean Diet; Microbioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet group (Experimental)
  Interventions: Dietary Supplement: Mediterranean Diet weaning scheme
- Control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Mediterranean Diet weaning scheme — Kids in experimental group were weaned by using fresh foods traditionally used in MD and appropriately adapted to infants including seasonal fruit and vegetables, various kinds of fresh blue fish, spices and herbs. No salt was used while a small amount of Parmesan cheese was added. No sugar was added to any meal.
  Arms: Mediterranean Diet group

SUMMARY:
A Randomized Controlled Clinical Trials was conducted to study the medium-long term impact of a complementary weaning using adult foods typical of Mediterranean Diets (MD) on children taste development and eating habits, and on the microbiota composition.

Main objectives were to assess the effect of such weaning scheme on:

1. medium-long term adherence of the children to the MD (Primary aim).
2. familial eating habits to verify how many changes may come from an early education of the kid toward a Mediterranean eating style
3. the BMI of the children
4. gut microbiota composition

ELIGIBILITY:
Inclusion Criteria:

* Infants, either breast fed or formula fed between 4 and 6 months of age
* Informed consent from at least one parent

Exclusion Criteria:

* Infants either with associated comorbidities or with low birth weight

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 394 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Proportions of children showing a good adherence (i.e. KidMed score >= 8) to Mediterranean diet | 36 months
  KidMed is a questionnaire measuring Mediterranean Diet Quality for children and adolescents. The final score ranges from from 0 to 12 where scores >=8 indicates optimal Mediterranean diet; score within range 4-7 suggest that an improvement is needed to adjust intake to Mediterranean patterns and score <=3 indicate very low diet quality.

SECONDARY OUTCOMES:
Average of the KidMed score | 36 months
Average children's BMI | 36 months
Proportion of overweight and obese children | 36 months
  Overweight and obesity were defined according to extra-centiles of the Italian BMI growth norms published in Cacciari et al. 2006.
Variation of microbial communities between arms based on Bray-Curtis dissimilarity | 48 months
  Bray-Curtis dissimilarity estimates difference in microbial abundances between two samples. It ranges from 0 to 1. The greater the index value the larger the difference in species abundances between groups.

REFERENCES:
- [Derived] de Franchis R, Bozza L, Cortese P, D'Antonio L, D'Avino A, Gasparini N, Ippolito G, Spadaro R, Tedesco M, Antignani A, De Filippis F, Valentino V, Auricchio R, Auricchio S, Bruzzese D. Can Early Nutrition Be Responsible for Future Gut Microbiota Changes and Different Health Outcomes? Nutrients. 2025 Nov 27;17(23):3721. doi: 10.3390/nu17233721. PMID 41374011